CLINICAL TRIAL: NCT05732155
Title: Preliminary Effectiveness of Individual and Group MDMA-assisted Therapy for Israeli Veterans With PTSD and Moral Injury From Special Forces Undercover Units
Brief Title: Preliminary Effectiveness of Individual and Group MDMA-assisted Therapy for Israeli Veterans With PTSD and Moral Injury.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: MAPS Public Benefit Corporation (MAPS PBC) 3141 Stevens Creek Blvd, #40547 San Jose, CA 95117 USA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC 00077-21
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder; Moral Injury; MDMA ('Ecstasy')
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Open-label study assesses the safety and preliminary effectiveness of MDMA-assisted therapy in participants diagnosed with PTSD. The study will be conducted in at least 30 participants. A flexible dose of MDMA HCl followed by a supplemental half dose unless tolerability issues emerge or a participant declines, is administered during the Treatment Period with manualized therapy in three open-label monthly Experimental Sessions (2 Experimental Individual Sessions, and one Experimental Group Session). This ~18-week Treatment Period is preceded by three Preparatory Sessions. Each Individual Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy. The Group Experimental Session is preceded by 2 Preparatory Group Sessions and followed by 3 Group Integrative Sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: methylenedioxymethamphetamine — The overall objective of this study is to use standard clinical measures to explore the safety and preliminary effectiveness of open-label MDMA-assisted therapy with a flexible dose of MDMA HCl, in participants with PTSD and moral injury, in individual and group treatment settings
  Other Names: group therapy model

SUMMARY:
The overall objective of this study is to use standard clinical measures to explore the safety and preliminary effectiveness of open-label MDMA-assisted therapy with a flexible dose of methylenedioxymethamphetaminel, in participants with Post traumatic Stress Disorder and moral injury, in individual and group treatment settings.

The overall safety objective is to assess the severity, incidence, and frequency of AEs, AEs of Special Interest (AESIs), and Serious Adverse Events (SAEs), concomitant medication use, suicidal ideation and behavior and vital signs .

DETAILED DESCRIPTION:
This single-site, open-label study assesses the safety and preliminary effectiveness of MDMA-assisted therapy in participants diagnosed with PTSD. All therapy teams have been trained by MAPS PBC. The study will be conducted in at least 30 participants. A flexible dose of MDMA HCl followed by a supplemental half dose unless tolerability issues emerge or a participant declines, is administered during the Treatment Period with manualized therapy in three open-label monthly Experimental Sessions (2 Experimental Individual Sessions, and one Experimental Group Session). This ~18-week Treatment Period is preceded by three Preparatory Sessions. Each Individual Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy. The Group Experimental Session is preceded by 2 Preparatory Group Sessions and followed by 3 Group Integrative Sessions. Experimental Sessions are followed by an overnight stay. The Primary Outcome measure, the change in PCL-5 from Baseline (Screening) will be repeated after each Experimental Session, with the final outcome assessed at ~35-weeks post Baseline (V18).

For each participant, the study will consist of:

* Screening Period: phone screen, informed consent, eligibility assessment, and Baseline assessments and enrollment of eligible participants
* Preparatory Period: medication tapering, Preparatory Sessions
* Treatment Period: three monthly Experimental Sessions and associated Integrative Sessions over ~17 weeks
* Follow-up Period and Study Termination: 1 week with no study visits, followed by Primary Outcome and Study Termination visit

After the Screening Period and Enrollment, eligible participants will begin a ~4-week Preparatory Period. Participants will attend three, 90-minute, non-drug, Preparatory Sessions (V1-3). Following the Preparatory Period, each participant will begin a ~17-week Treatment Period consisting of an Individual phase and a Group phase, with 2 Individual Experimental Sessions, and 1 Group Experimental Session. The Individual Experimental Sessions will each be followed by three Individual Integrative Sessions, and the Group Experimental Session will be followed by two Group Integrative Sessions. MDMA will be administered three times during the Treatment Period (V4, V8, and V14). The Experimental Sessions will last ~8 hours. Three 90-minute Individual Integration Sessions and a PCL-5 assessment (as an exploratory measure) will follow the first and second Individual Experimental Session (V4 and V8), each a week apart. The first Individual Integration Session (V5) will occur the morning following V4, and the next Individual Integration Session (V6) will occur a week later. The PCL-5 (V7) is administered a week after V6, at the third Integration Session (V7). The same regimen will follow Treatment 2 (V8): an Individual Integration Session (V9) will occur the morning following V8, the next Individual Integration Session (V11) a week later, PCL-5 assessment will take place at the same visit of the third Integration Session (V11) one week later. Finally, the Group treatment period will begin 2-10 weeks after V11. n order to synchronize between all individual participants, after their different dates completing V11, and to allow their joint synchronized commencement of the group phase. To reduce this time variability to a minimum, the Individual group members will commence their Individual treatment period within the same week as the rest of the group. Since the study team must recruit and screen potentially eligible participants (see Section 5.6 Recruitment Strategies), coordinate schedules among participating staff members, and coordinate medication taper plans and assessments there must be adequate flexibility factored into the timing of screening, initial enrollment, and scheduling. The timing of initial enrollment for participants may be delayed or adjusted at the sponsor-investigator's discretion. The group phase will begin with two 90-minute Preparatory Sessions (V12-V13), focused on enabling acquaintance among group members, and discussing the individual goals of each group member. Three Integration Sessions (V15-17), each a week apart, will follow the third Experimental Group Session (V14). V15 will take place the morning after V14. The Primary Outcome measure will be the change in PCL-5 Score from Screening (Baseline) to V18 (Outcome), ~7 weeks after the final Experimental Session (V14) and ~4 weeks after the final Integration Session (V17), and assessed by a rater from the research team. V18 will also be the study termination visit.

ELIGIBILITY:
Inclusion Criteria:

* Are veterans of special forces undercover units in the Israeli army.
* Are fluent in speaking and reading the predominantly used or recognized language of the study site (Hebrew).
* Are able to swallow pills.
* Agree to have study visits recorded, including Experimental Sessions, and non-drug psychotherapy sessions.
* Must provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* Agree to the following lifestyle modifications : comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not participate in any other interventional clinical trials during the duration of the study, remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures.
* At Screening, meet DSM-5 criteria for current PTSD with a symptom duration of 6 months or longer.
* At Screening, have at least moderate PTSD symptoms in the last month, based on PCL-5 total score of 36 or greater.
* May have well-controlled hypertension.
* May have asymptomatic Hepatitis C virus (HCV).
* May have alcohol or substance use disorder.
* May have a history of or current Diabetes Mellitus (Type 2).
* May have hypothyroidism if taking adequate and stable thyroid replacement medication.
* May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial.
* Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the sponsor-investigator or study clinician, contraindicates participation in the study.
* Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
* Have a history of or a current primary psychotic disorder.
* Have a current eating disorder with active purging assessed via MINI and clinical interview.
* Have current major depressive disorder with psychotic features assessed via MINI.
* Have a current alcohol or substance use disorder other than caffeine or nicotine that the investigators, therapy team, and/or study physician judge to be a safety concern for enrollment in the study.
* Have an active illicit (other than cannabis) or prescription drug substance use disorder at any severity within 12 months prior to enrollment.
* Have current Personality Disorders.
* .Any participant presenting current serious suicide risk,
* Require ongoing concomitant therapy with a psychiatric medication with exceptions described in protocol section on Concomitant Medications.
* Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate.
* Have uncontrolled essential hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions).
* Have a history of ventricular arrhythmia at any time, other than premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
* Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
* Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.
* Have a marked Baseline prolongation of QT/QTc interval . QTc interval > 450 milliseconds (ms) in males and >460 ms in females corrected using Fridericia's formula.
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions.
* Have symptomatic liver disease or have significant liver enzyme elevations.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Have engaged in ketamine-assisted therapy or used ketamine within 12 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the change in PCL-5 (PTSD Checklist for DSM-5 ) from Baseline | Maximum 46 weeks
  The primary endpoint is the change in mean PCL-5 Scores from Baseline (T1, Screening) to Primary Outcome Visit (T5, V18). Analysis of the primary endpoint will be conducted using an ANCOVA model, comparing PCL-5 scores at baseline and at primary endpoint, while adjusting for baseline PCL-5 and potential covariates. The primary endpoint analyses will be based on the mITT analysis set plus DSP4. Adjustment for additional potential covariates and subgroups will be explored. Additional details will be provided in the SAP.

IPD SHARING:
Plan to Share IPD: No
Participants will be assigned a unique identifier by the sponsor-investigator. Any participant records or datasets that are transferred will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.